CLINICAL TRIAL: NCT03396120
Title: The FVC/DLCO Ratio is a Useful Predictor of Pulmonary Hypertension in Patients With Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU6
Record Dates: First submitted 2018-01-05; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Interstitial Lung Disease; Pulmonary Hypertension
MeSH Terms: conditions — Lung Diseases, Interstitial; Hypertension, Pulmonary | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pulmonary function test — forced vital capacity and diffusing capacity
  Other Names: FVC/DLCO

SUMMARY:
Pulmonary hypertension (PH) is a common disorder among patients with interstitial lung disease (ILD). The symptoms are usually nonspecific and overlooked. Thus, a noninvasive screening modality is recommended for early detection of PH because of its potentially significant impact on treatment strategy and clinical outcomes.

Objectives: To evaluate the usefulness of assessing forced vital capacity (FVC%), diffusion capacity of the lung for carbon monoxide (DLCO%), and FVC%/DLCO% ratio to predict pulmonary hypertension among patients with ILDs.

ELIGIBILITY:
Inclusion Criteria:

* This retrospective study included all patients diagnosed with interstitial lung disease (ILD) who were followed up by the chest department of a tertiary hospital between September 2016 and January 2017

Exclusion Criteria:

* patients with occupational history
* collagen vascular disease predisposing them to lung disorders
* patients who could not undergo pulmonary function testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - ILD was diagnosed on the basis of clinical, radiological and functional assessments
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
value of FVC/DLCO in predicting PAH in IPF | 6 months
  To evaluate the usefulness of assessing forced vital capacity (FVC%), diffusion capacity of the lung for carbon monoxide (DLCO%), and FVC%/DLCO% ratio to predict pulmonary hypertension among patients with ILDs

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - AssiutU, Asyut
  - Pulmonology Departments, Asyut

IPD SHARING:
Plan to Share IPD: No